CLINICAL TRIAL: NCT02452658
Title: Detecting Changes on Fast Food Menu
Brief Title: Fast Food Photo Study 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carnegie Mellon University (Other)
Responsible Party: Principal Investigator, Eric VanEpps, PhD Candidate, Carnegie Mellon University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HS14-582 Study 2
Record Dates: First submitted 2015-05-19; First posted 2015-05-22 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Obesity
Keywords: Fast food literacy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Changed menu (Experimental): All participants will be exposed to the same changed menu after making their hypothetical choice. Changes will include reduced calorie labels, reduced prices, and changes to item descriptions.
  Interventions: Other: Changed menu

INTERVENTIONS:
Other: Changed menu — After making the hypothetical choice, participants will be exposed to a menu with changed calorie and price labels, as well as several other changes.

SUMMARY:
Participants will be exposed to a hypothetical fast food menu, asked to place a hypothetical lunch order, and will then be exposed to a second menu with several changes made to the menu. Participants will be asked to identify as many changes as possible on this second menu, and then complete a survey about their eating tendencies and demographics.

DETAILED DESCRIPTION:
The menu with changes will feature changes to both calories and prices, allowing for measures of whether participants notice such changes and the order in which changes are noticed.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older,
* agrees to consent form

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 311 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of participants who notice calorie change | Participants will have 2 minutes to notice changes on the menu
Number of participants who notice price change | Participants will have 2 minutes to notice changes on the menu

SECONDARY OUTCOMES:
Within-participant ranking of the order in which changes were noticed | Participants will have 2 minutes to notice changes on the menu
Total number of changes noticed | Participants will have 2 minutes to notice changes on the menu

CONTACTS AND LOCATIONS:
Overall Officials: Eric M VanEpps, PhD, Principal Investigator — Graduated PhD Candidate
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States